CLINICAL TRIAL: NCT02374099
Title: A Phase 2, Randomized, Open-label, Two-arm Study to Assess the Efficacy and Safety of the Epigenetic Modifying Effects of CC-486 (Oral Azacitidine) in Combination With Fulvestrant in Postmenopausal Women With ER+, HER2- Metastatic Breast Cancer Who Have Progressed on an Aromatase Inhibitor
Brief Title: Study to Assess the Efficacy and Safety of the Epigenetic Modifying Effects of CC-486 (Oral Azacitidine) in Combination With Fulvestrant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-486-BRSTM-001
Expanded Access: NCT03723135 (Approved for marketing)
Record Dates: First submitted 2015-01-22; First posted 2015-02-27 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Her2 -; ER+; CC-486 (ORAL AZACITIDINE); Metastatic Breast Cancer; Oral Azacitidine; Fulvestrant; Epigenetics
MeSH Terms: conditions — Breast Neoplasms | interventions — cc-486; Azacitidine; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CC-486 and fulvestrant (Experimental): CC-486 300 mg by mouth (PO) daily on days 1-21 of each 28 day cycle and fulvestrant 500mg by intramuscular (IM) injection on Days 1 and 15 of cycle 1 and day 1 of each subsequent cycle every 28 days.
  Interventions: Drug: CC-486; Drug: Fulvestrant
- Fulvestrant (Experimental): Fulvestrant will be administered by intramuscular injection at a dose of 500 mg on days 1 and 15 of cycle 1 and day 1 of subsequent cycles.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: CC-486 — Each cycle will be 28 days. CC-486 will be administered orally at a dose of 300 mg daily on days 1-21 of each 28-day cycle
  Other Names: Oral Azacitidine
  Arms: CC-486 and fulvestrant
Drug: Fulvestrant — Fulvestrant will be administered by intramuscular (IM) injection at a dose of 500 mg on days 1 and 15 of cycle 1 and day 1 of subsequent cycles.
  Other Names: Faslodex

SUMMARY:
The purpose of this study to Assess the Efficacy and Safety of the Epigenetic Modifying Effects of CC-486 (Oral Azacitidine) in Combination With Fulvestrant in Postmenopausal Women with estrogen receptor positive (ER+), human epidermal growth factor receptor 2 (HER2-) Metastatic Breast Cancer Who Have Progressed on an Aromatase Inhibitor (AI).

DETAILED DESCRIPTION:
This is a Phase 2, open-label, two-arm study assessing the efficacy and safety of the combination of fulvestrant with CC-486 in subjects with ER+, HER2- metastatic breast cancer who have progressed after prior AI.

Approximately 92 participants will be enrolled and assigned randomly in a 1:1 ratio to one of two treatment arms:

* Arm A: CC-486 300 mg and fulvestrant 500 mg: 46 subjects
* Arm B: Fulvestrant 500 mg: 46 subjects Each cycle will be 28 days. CC-486 will be administered orally at a dose of 300 mg daily on days 1-21 of each 28-day cycle. Fulvestrant will be administered by intramuscular (IM) injection at a dose of 500 mg on days 1 and 15 of cycle 1 and day 1 of subsequent cycles.

Safety will be evaluated by an independent data monitoring committee (DMC) after a total of approximately 32 subjects have completed at least 1 treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female ≥ 18 years of age (at the time of signing the informed consent form) with metastatic breast cancer not amenable to curative treatment by surgery or radiotherapy.
* Subject is considered postmenopausal
* Subject has a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive breast cancer by local laboratory (based on most recently analyzed biopsy).
* Subject has human epidermal growth factor receptor 2 negative (HER2-) breast cancer (based on most recently analyzed biopsy) defined as a negative in situ hybridization test or an Immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing.
* Subject had disease refractory to an AI
* Subject has an Eastern Cooperative Oncology Group ( ECOG) performance status of 0-1.
* Subject has radiological documented measurable disease (ie, at least one measureable lesion as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1).

  * If no measurable disease is present, then at least one predominantly lytic bone lesion must be present
* Subject has adequate organ function.
* Subject has adequate bone marrow function.

Exclusion Criteria:

* Subject has received > 1 prior line of chemotherapy in the metastatic setting
* Subject has received any chemotherapy within 21 days prior to randomization.
* Subject has received prior treatment with fulvestrant.
* Subject has been previously treated with azacitidine (any formulation), decitabine, or any other hypomethylating agent.
* Subject has a history of, or current symptomatic brain metastasis.
* Subject has severe renal impairment (creatinine clearance < 30 ml/min).
* Subject has an impaired ability to swallow oral medication.
* Subject has a contraindication to receiving IM injections (eg, bleeding disorders, anticoagulant use).
* Subject has significant active cardiac disease within the previous 6 months including unstable angina or angina requiring surgical or medical intervention, significant cardiac arrhythmia, or New York Heart Association (NYHA) class 3 or 4 congestive heart failure.
* Subject is a female of Childbearing Potential [defined as a sexually mature woman who (1) has not undergone hysterectomy (the surgical removal of the uterus) or bilateral oopherectomy (the surgical removal of both ovaries) or (2) has not been naturally postmenopausal for at least 12 consecutive months (ie, has had menses at any time during the preceding 12 consecutive months)].

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-03-13 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ileana Elias, MD, Study Director — Celgene
Locations (35):
- United States (8):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - Virginia G Piper Cancer Center, Scottsdale, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Florida Cancer Specialists, West Palm Beach, Florida
  - University of Kansas Hospital, Westwood, Kansas
  - Henry Ford Health System, Detroit, Michigan
  - Clinical Research Alliance, New York, New York
  - Medical Oncology Associates, Spokane, Washington
- Belgium (4):
  - Grand Hopital de Charleroi, Charleroi
  - AZ Groeninge, Kortrijk
  - Clinique Sainte Elisabeth - Service d'Oncologie, Namur
  - GasthuisZusters Antwerpen, Wilrijk
- France (4):
  - Centre Regional de lutte contre le cancer Paul Papin, Angers
  - Institut Bergonie, Borddeaux Cedex
  - Hopital Pitie Salpetriere, Paris
  - Centre Rene Gauducheau Centre de Lutte Contre Le Cancer Nantes Atlantique, Saint-Herblain
- Germany (4):
  - Universitatsklinikum Hamburg-Eppendorf / IVDP, Hamburg
  - Hamatologisch Onkologische Praxis Eppendorf, Hamburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - TU München - Klinikum rechts der Isar, München
- Italy (8):
  - Policlinico S. Orsola - Malpighi, Bologna
  - Ospedale San Raffaele S.r.l., Milan
  - Istituto Nazionale Dei Tumori, Milan
  - IEO- Istituto Europeo di Oncologia, Milan
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Policlinico Umberto I, Roma
  - Policlinico Universitario A Gemelli, Roma
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino, Piemonte
- Spain (7):
  - Complejo Universitario La Coruna, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall D Hebron, Barcelona
  - Hospital General Gregorio Maranon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico Universitario Virgen de La Victoria, Málaga
  - Hospital Virgen del Rocio, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 35 sites in Spain, Germany, Belgium, Italy and the United States.
Pre-assignment Details: The study enrolled adult, postmenopausal women, with metastatic breast cancer who progressed on an aromatase inhibitor. Participants were randomly assigned in a 1:1 ratio to one of two treatment arms to CC-486 tablets and fulvestrant or fulvestrant alone.
Groups:
- CC-486 and Fulvestrant: Participants received CC-486 tablets by mouth (PO) daily (QD) on days 1-21 of each 28 day treatment cycle and fulvestrant 500 mg by intramuscular injection (IM) on days 1 and 15 of cycle 1 and on day 1 only in subsequent cycles until disease progression, start of new anticancer therapy, death, withdrawal of consent, or lost to follow-up withdrawal of consent, or lost to follow-up.
- Fulvestrant: Participants received fulvestrant 500 mg by intramuscular injection on days 1 and 15 of cycle 1 and on day 1 only in subsequent cycles until disease progression, start of new anticancer therapy, death, withdrawal of consent, or lost to follow-up.
Period: Overall Study
Arm/Group | CC-486 and Fulvestrant | Fulvestrant
Started | 48 | 49
Participants Treated | 46 (2 participants randomized, but not treated) | 48 (1 participant randomized, but not treated)
Completed | 0 | 0
Not Completed | 48 | 49
Not completed — Adverse Event | 1 | 0
Not completed — Progressive Disease | 35 | 40
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Miscellaneous | 2 | 3
Not completed — Randomized, but not treated | 2 | 1
Not completed — Study Terminated by Sponsor | 3 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population includes all randomized participants regardless of whether the participant received any investigational product (IP) or had any efficacy assessments collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | CC-486 and Fulvestrant | Fulvestrant | Total
Number analyzed (Participants) | 48 | 49 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.99) | 62.9 (10.03) | 62.7 (10.46)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 29 | 25 | 54
  From 65-84 years | 19 | 24 | 43
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 0 | 0 | 0
Race [Count of Participants; unit: Participants]
  White | 34 | 39 | 73
  Asian | 0 | 1 | 1
  American Indian/Alaska Native | 1 | 0 | 1
  Not Collected or Reported | 13 | 9 | 22
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a subject's disease is progressing, assess how the disease affects the daily living activities of the subject and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = Fully Active | 36 | 21 | 57
    1 = Restrictive but ambulatory | 12 | 28 | 40
    2 = = Ambulatory but unable to work | 0 | 0 | 0
    3 = Limited Self Care | 0 | 0 | 0
Histology of Primary Diagnosis [Number; unit: Participants]
  Ductal (Scirrhous Carcinoma) | 37 | 38 | 75
  Lobular Carcinoma | 7 | 12 | 19
  Other, Not specified | 4 | 2 | 6
  Missing | 2 | 1 | 3
Time from Primary Diagnosis of Breast Cancer to Study Randomization [Mean (Standard Deviation); unit: months] | 119.05 (70.322) | 95.57 (76.434) | 107.19 (74.037)
Duration of Prior Hormonal Anti-Cancer Therapy [Mean (Standard Deviation); unit: Months] | 31.39 (14.830) | 35.84 (27.409) | 33.64 (22.097)

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Progression Free Survival (PFS)
Description: Progression-free survival was defined as the duration from the date of randomization to the date of disease progression (DP) based on investigator's assessment using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 or death (from any cause), whichever occurred first. Per RECIST 1.1, progressive disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions from nadir or appearance of a new lesion.
Time Frame: From the date of randomization of study drug to the date of the cut off date of 13 December 2016; follow-up for PFS was 21 months
Population: The Intent-to-treat population included all randomized participants regardless of whether the participant received any investigational product or had any efficacy assessments collected.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CC-486 and Fulvestrant | Fulvestrant
Number analyzed (Participants) | 48 | 49
months | 5.49 [2.07 to 8.25] | 5.46 [3.58 to 7.36]
Statistical Analysis 1: Comparison: CC-486 and Fulvestrant vs Fulvestrant; Test type: Superiority; p = 0.599, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.54 to 1.42]; Hazard ratio and associated two-sided 95% confidence intervals (CI) were estimated by the Cox proportional hazard models

2. Secondary Outcome: Percentage of Participants Who Achieved a Confirmed Complete Response (CR) or Partial Response (PR) to Treatment (Objective Response Rate) Based On the Investigator Assessment
Description: Overall response rate was defined as the percentage of participants who achieved a confirmed complete response or partial response based on RECIST Version 1.1 criteria. RECIST criteria v 1.1 defined a CR as the disappearance of all target lesions and a PR with at least a 30% decrease in the sum of diameters of target lesions from baseline. The two-sided 95% exact binomial CI for each arm was estimated by the Clopper-Pearson method.
Time Frame: Disease response was assessed every 8 weeks, for the first 24 weeks, then every 12 weeks until DP; from date of randomization of study drug to data cut-off date of 13 December 2016; follow-up for overall response was 21 months
Population: The ITT population included all randomized participants regardless of whether the participant received any IP or had any efficacy assessments collected.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CC-486 and Fulvestrant | Fulvestrant
Number analyzed (Participants) | 48 | 49
Percentage of Participants | 8.3 (2.32) [2.32 to 19.98] | 2.0 (0.05) [0.05 to 10.85]
Statistical Analysis 1: Comparison: CC-486 and Fulvestrant vs Fulvestrant; Test type: Superiority; p = 0.1479, Fisher Exact; Difference in Response Rates = 6.3, 95% CI 2-sided [-2.47 to 15.06]; The two-sided 95% confidence interval for the difference in ORR was estimated by the Wilson method

3. Secondary Outcome: Percentage of Participants Who Achieved a Confirmed CR, PR or Stable Disease (SD) for ≥ 24 Weeks (Clinical Benefit Rate) by Investigator Assessment
Description: Percentage of participants with CR or PR or SD was defined per RECIST criteria v 1.1 as a CR that includes a disappearance of all target lesions, a PR was defined as having at least a 30% decrease in the sum of diameters of target lesions from baseline and SD as neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for progressive disease. The two-sided 95% exact binomial CI each arm was estimated by the Clopper-Pearson method.
Time Frame: Disease response was assessed every 8 weeks, for the first 24 weeks, then every 12 weeks until DP; from date of randomization of study drug to the data cut-off date of 13 December 2016; follow-up for clinical benefit response was 21 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CC-486 and Fulvestrant | Fulvestrant
Number analyzed (Participants) | 48 | 49
Percentage of Participants | 31.3 (18.66) [18.66 to 46.25] | 30.6 (18.25) [18.25 to 45.42]
Statistical Analysis 1: Comparison: CC-486 and Fulvestrant vs Fulvestrant; Test type: Superiority; p = 0.1732, Fisher Exact; Difference in Clinical Benefit Rate = 0.7, 95% CI 2-sided [-17.76 to 19.04]; The two-sided 95% confidence interval for the difference in clinical benefit rate was estimated by the Wilson method

4. Secondary Outcome: Kaplan Meier Estimate of Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death (from any cause). All participants who were lost to follow up prior to the end of the study or who were withdrawn from the study were censored at the time of last contact.
Time Frame: From the date of randomization of study drug to the data cut off date of 13 December 2016; participants were followed for overall survival for 21 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CC-486 and Fulvestrant | Fulvestrant
Number analyzed (Participants) | 48 | 49
months | NA [13.7 to NA] — NA = indicates overall survival was not estimable due to the insufficient number of participants with events at the time of the cut-off date. The median OS was not reached. | NA [10.7 to NA] — NA = indicates overall survival was not estimable due to the insufficient number of participants with events at the time of the cut-off date. The median OS was not reached.
Statistical Analysis 1: Comparison: CC-486 and Fulvestrant vs Fulvestrant; Test type: Superiority; p = 0.2725, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.23 to 1.53]; Hazard Ratio and associated two-sided 95% CI were estimated by the Cox proportional hazard model

5. Secondary Outcome: Kaplan Meier Estimate of Duration of Response (DoR)
Description: Duration of response was defined as the time from the first tumor assessment when the confirmed CR/PR criterion was first met to the date of disease progression, based on investigator's assessment following RECIST Version 1.1 criteria.
Time Frame: From the date of randomization of study drug to the data cut-off of 13 December 2016; follow up for duration of response was 21 months
Population: Only participants who had a confirmed CR or PR response are included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CC-486 and Fulvestrant | Fulvestrant
Number analyzed (Participants) | 48 | 49
months | NA [6.61 to NA] — NA = indicates duration of response was not estimable due to the data not being mature at the time of the data cut off date. The median DOR was not reached. | NA [NA to NA] — NA = indicates duration of response was not estimable due to the data not being mature at the time of the data cut off date. The median DOR was not reached.

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events (TEAEs) were defined as any AEs that begin or worsen with an onset date on or after the date of the first dose of IP through 28 days after the last dose. A serious AE (SAE) = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs were graded based on the participant's symptoms according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0); AEs were evaluated for severity as follows: Grade 1 = Mild - transient or mild discomfort; no medical intervention required; Grade 2 = Moderate - mild to moderate limitation in activity; Grade 3 = Severe; Grade 4 = Life threatening; Grade 5 = Death.
Time Frame: Randomization to 28 days after the last dose of IP; those AEs known at any time thereafter being related to IP; up to the last subject last visit of 21 November 2017; TEAE follow-up occurred up to 155 weeks and 2 days
Population: The safety population included all randomized participants who received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | CC-486 and Fulvestrant | Fulvestrant
Number analyzed (Participants) | 46 | 48
Participants
  TEAE | 46 | 45
  Grade 3 or 4 TEAE | 32 | 15
  Grade 5 TEAE (Death) | 2 | 1
  Serious TEAE | 10 | 7
  TEAE Leading to Stopping of Any IP | 14 | 1
  TEAE Leading to Dose Reduction of any IP | 19 | 0
  TEAE Leading to Dose Interruption of any IP | 22 | 3
  Treatment Related TEAE | 46 | 31
  Treatment Related TEAE Grade 3 or 4 TEAE | 29 | 2
  Treatment Related TEAE Grade 5 Death | 0 | 0
  Treatment Related Serious TEAE | 4 | 0

ADVERSE EVENTS:
Time Frame: From randomization date to 28 days after the last dose of IP; those AEs known at any time thereafter being related to IP; up to last subject last visit date of 21 November 2017.
Arm/Group | CC-486 and Fulvestrant | Fulvestrant
All-Cause Mortality (participants affected / at risk) | 14/46 | 16/48
Serious Adverse Events (participants affected / at risk) | 10/46 | 7/48
Other Adverse Events (participants affected / at risk) | 45/46 | 44/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-486 and Fulvestrant (N=46) | Fulvestrant (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC-486 and Fulvestrant (N=46) | Fulvestrant (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 10 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 19 | 10
Diarrhoea (Gastrointestinal disorders) | 20 | 6
Nausea (Gastrointestinal disorders) | 35 | 14
Vomiting (Gastrointestinal disorders) | 33 | 5
Asthenia (General disorders) | 16 | 10
Fatigue (General disorders) | 13 | 12
Injection site pain (General disorders) | 1 | 5
Oedema peripheral (General disorders) | 1 | 3
Pyrexia (General disorders) | 3 | 2
Urinary tract infection (Infections and infestations) | 3 | 4
Viral upper respiratory tract infection (Infections and infestations) | 3 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 5
Blood alkaline phosphatase increased (Investigations) | 0 | 3
Weight decreased (Investigations) | 3 | 1
White blood cell count decreased (Investigations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 13 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 6
Dizziness (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 5 | 5
Anxiety (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Hot flush (Vascular disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.